CLINICAL TRIAL: NCT02003339
Title: Pilot Prospective Study on Interest of Functional MRI in Early Assessment of Radioembolization Efficiency in Patients Suffering From Hepatocellular Carcinoma
Brief Title: Interest of Functional MRI (Magnetic Resonance Imagery) (in Patients Suffering From Hepatocellular Carcinoma and Treated With Yttrium
Acronym: ICY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-JE-CHC-Pron; 2012-A00972-41 (Registry Identifier: ANSM)
Record Dates: First submitted 2013-11-25; First posted 2013-12-06 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RMIs (Experimental)
  Interventions: Other: Additional RMIs

INTERVENTIONS:
Other: Additional RMIs

SUMMARY:
For patients who are suffering from hepatocellular carcinoma and are treated with radioembolization, the purpose of this study is to analyse parameters of functional MRIs that are modified early and to detect parameters that vary significantly after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Early, intermediate, advanced, non metastatic Hepatocellular Carcinoma. Indication for radioembolization validated after pluridisciplinary committee meeting.
* Isolated target on initial imagery (invasive hepatocellular carcinoma excluded)
* WHO (World Health organization) Performance status: 0, 1 or 2
* If cirrhosis, Child A score with total bilirubin less than 30 micromoles per liter
* Creatinine clearance more or equal to 30 mL/min
* Patient informed and consent signature obtained

Exclusion Criteria:

* Invasive hepatocellular carcinoma without any isolated tumor
* Disease needing 2 injections of Therasphere
* Thrombosis extending into the porta(thrombosis of one of left or right branch authorized), extra hepatic metastasis
* Previous treatment by chemoembolization, radiofrequency less than 3 months before radioembolization
* No antiangiogenic concomitant treatment, 15 days before and 15 days after radioembolization, including Sorafenib
* Associated disease which could prevent patient from receiving treatment
* RMI contre-indication(particle or metal prosthesis, pacemaker, claustrophobia) or contrast product contre-indication (allergy)
* Patient already participating in an other therapeutic trial with an experimental drug
* Pregnant or childbearing potential women or breastfeeding women
* minors, persons deprived of liberty or protected adults (maintenance of justice, guardianship or supervision) Unable to comply with trial medical follow-up for geographical, social or psychological reasons
* Unable to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Modifications of functional MRI parameters | Before radioembolization and up to 6 months after radioembolization

SECONDARY OUTCOMES:
Correlation between functional MRIs parameters and tumoral response | Measured 6 months after radioembolization
Assessment of alternative morphological response criteria : EASL (European Association for study of the liver) and mRECIST (m response evaluation criteria in solid tumor) criteria. Link with RECIST response. | 2 and 6 months
Change of VEGF (vascular endothelial growth factor) release | From day 0 to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien EDELINE, MD, Principal Investigator — Centre Eugène Marquis
Locations (1):
- Centre Eugène Marquis, Rennes, France